CLINICAL TRIAL: NCT07369401
Title: Efficacy and Safety of Deep Brain Stimulation of the Nucleus Accumbens and Anterior Limb of the Internal Capsule in the Treatment of Refractory Schizophrenia: A Prospective, Single-Center, Double-Blind, Randomized Controlled Study
Brief Title: Deep Brain Stimulation of the Nucleus Accumbens and Anterior Limb of the Internal Capsule in the Treatment of Refractory Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, De-zhi Kang, professor, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRCTA,ECFAH of FMU [2025]637
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Refractory Schizophrenia
Keywords: Deep Brain Stimulation; Refractory Schizophrenia; Nucleus Accumbens; Anterior Limb
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessing physicians are blinded, while programming physicians are unblinded. Initial stimulation parameters are 2.5-7.5 V, 60-210 μs, and 80-210 Hz. During the stabilization phase, parameters are adjusted individually in the order of "voltage → pulse width/frequency → contacts/mode", and patients are not informed of adjustments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group 1 (Experimental): DBS is activated 2 weeks after implantation for NAcc-only stimulation. Stimulation is maintained for 6 weeks (until week 8 postoperatively), then shut down. Stimulation is reactivated at week 10 for anterior limb of the internal capsule-only stimulation, maintained for 6 weeks (until week 16 postoperatively), then shut down. Combined stimulation of the NAcc and anterior limb of the internal capsule is initiated at week 18 postoperatively, maintained for 6 weeks, followed by efficacy assessment.
  Interventions: Device: Deep Brain Stimulation
- Trial Group 2 (Experimental): DBS is activated 2 weeks after implantation for anterior limb of the internal capsule-only stimulation. Stimulation is maintained for 6 weeks (until week 8 postoperatively), then shut down. Stimulation is reactivated at week 10 for NAcc-only stimulation, maintained for 6 weeks (until week 16 postoperatively), then shut down. Combined stimulation of the NAcc and anterior limb of the internal capsule is initiated at week 18 postoperatively, maintained for 6 weeks, followed by efficacy assessment.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — An assessment is conducted 7 days postoperatively. DBS is activated 2 weeks after implantation for NAcc-only stimulation. Stimulation is maintained for 6 weeks (until week 8 postoperatively), then shut down. Stimulation is reactivated at week 10 for anterior limb of the internal capsule-only stimulation, maintained for 6 weeks (until week 16 postoperatively), then shut down. Based on the participant's vital signs and motor responses to stimulation, initial parameters are set as: 2.5-7.5 V, pulse width 60-210 µs, frequency 80-210 Hz. During the stabilization phase, an independent clinical programmer adjusts parameters individually for each patient based on clinical status and provides guidance according to symptom changes. Patients are not informed of any adjustments. To maximize therapeutic efficacy, the adjustment sequence is: (1) increase voltage up to 7.5 V; (2) increase pulse width or frequency up to 210 µs/Hz; (3) change contacts or modes (monopolar negative or bipolar negative).
  Arms: Trial Group 1
Device: Deep Brain Stimulation — An assessment is conducted 7 days postoperatively. DBS is activated 2 weeks after implantation for anterior limb of the internal capsule-only stimulation. Stimulation is maintained for 6 weeks (until week 8 postoperatively), then shut down. Stimulation is reactivated at week 10 for NAcc-only stimulation, maintained for 6 weeks (until week 16 postoperatively), then shut down.Based on the participant's vital signs and motor responses to stimulation, initial parameters are set as: 2.5-7.5 V, pulse width 60-210 µs, frequency 80-210 Hz. During the stabilization phase, an independent clinical programmer adjusts parameters individually for each patient based on clinical status and provides guidance according to symptom changes. Patients are not informed of any adjustments. To maximize therapeutic efficacy, the adjustment sequence is: (1) increase voltage up to 7.5 V; (2) increase pulse width or frequency up to 210 µs/Hz; (3) change contacts or modes (monopolar negative or bipolar negative).
  Arms: Trial Group 2

SUMMARY:
Schizophrenia is a lifelong psychiatric disorder with a prevalence rate of 0.559% and a lifetime prevalence rate of 0.588% among Chinese adults. It often causes social dysfunction and psychiatric disability, shortening patients' life expectancy by 10-25 years compared to the general population. Approximately 30% of patients are resistant to antipsychotic medications, and 60% of these do not respond to clozapine (ultra-refractory). DBS has shown definite efficacy in movement disorders and refractory obsessive-compulsive disorder (OCD) as well as major depressive disorder (MDD). Preliminary studies have indicated that DBS targeting sites such as the NAcc can improve symptoms in some schizophrenia patients. Additionally, abnormal white matter in the anterior limb of the internal capsule has been identified in refractory patients, providing a basis for exploring combined target stimulation.

This study aims to investigate the efficacy and safety of deep brain stimulation of the Nucleus Accumbens and Anterior Limb of the Internal Capsule in the treatment of refractory schizophrenia. A randomized controlled (self-controlled) design is adopted. The statistical analysis unit generates a random allocation table using SAS software, and groups are assigned via central randomization. Both groups undergo three stimulation phases: DBS activation 2 weeks after surgery, 6 weeks of single-target stimulation followed by 2 weeks of shutdown, another 6 weeks of alternate single-target stimulation followed by 2 weeks of shutdown, and finally 6 weeks of combined dual-target stimulation. Trial Group 1 is stimulated sequentially at NAcc, Anterior Limb of the Internal Capsule, and dual targets; Trial Group 2 follows the reverse order for single-target stimulation before combined stimulation. Surgery is performed under general anesthesia by neurosurgeons with associate senior titles or above and extensive experience. After head frame placement, CT and MRI images are fused for targeting. Electrodes are implanted into the NAcc via the Anterior Limb of the Internal Capsule, and a pulse generator is placed under the clavicle and connected to the electrodes. Postoperative CT confirms electrode position. Trial devices are provided by Jingyu Medical Technology (Suzhou) Co., Ltd., including implantable neurostimulation systems, electrode leads, extension leads, and programming equipment. On-site follow-up is conducted at key time points: screening, baseline, 2 weeks postoperatively (DBS activation), 6 weeks after stimulation, 16 weeks postoperatively, and 24 weeks postoperatively, including scale assessments, physical examinations, and laboratory/imaging tests. The primary outcome measure was the reduction rate of the total PANSS score at 24 weeks after DBS implantation compared to baseline, with a 20% reduction defined as effective, assessed by independent psychiatric evaluators.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years (inclusive) at the time of signing the informed consent form, male or non-pregnant female;
* Meets the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for schizophrenia;
* Schizophrenia disease course ≥ 5 years before screening;
* Meets the 2016 TRRIP criteria for refractory/ultra-refractory schizophrenia: previous treatment with ≥ 2 non-clozapine antipsychotics at adequate dose (≥ 600mg/day chlorpromazine equivalent) and duration (≥ 12 weeks) with no response or intolerance, or clozapine at adequate dose (≥ 300mg/day or plasma concentration ≥ 350ng/ml) and duration (≥ 12 weeks) with no response or intolerance, plus moderate or greater symptom severity;
* PANSS total score ≥ 70 at screening and baseline;
* No changes in medication regimen in the past 2 months;
* The patient and their guardian have been fully informed and signed the informed consent form.

Exclusion Criteria:

* Comorbid with epilepsy, severe cognitive impairment (Mini-Mental State Examination [MMSE] score < 10), organic mental disorder, paranoid personality disorder, mental retardation, or addiction (other than nicotine);
* Has implanted devices such as cochlear implants or cardiac pacemakers, or has undergone surgery that may affect the trial within 6 months;
* Has contraindications to DBS implantation and is deemed unsuitable for surgery by the investigator;
* Has participated in other drug/medical device clinical trials within 3 months before screening;
* Confirmed HIV-positive;
* Pregnant/lactating women, women of childbearing age with positive HCG/urine pregnancy test at screening, those unable to use effective contraception during the trial, or those planning to conceive within 3 months after trial initiation;
* Other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The reduction rate of the total PANSS score at 24 weeks | 24 weeks after treatment
  The reduction rate of the total PANSS score at 24 weeks after DBS implantation compared to baseline. The reduction rate is (PANSS score at baseline - PANSS score at 24-weeks) / PANSS score at baseline. PANSS score was assessed by independent psychiatric evaluators.

SECONDARY OUTCOMES:
The proportion of effective treatment | 24 weeks after treatment
  Compared with the baseline, a reduction of ≥ 20% in the total PANSS score is defined as effective treatment. The reduction rate is (PANSS score at baseline - PANSS score at 24-weeks) / PANSS score at baseline. PANSS score was assessed by independent psychiatric evaluators.
The change value of the Clinical Global Impression (CGI) scale score at 24 weeks | 24 weeks after treatment
  Changes in the Clinical Global Impression (CGI) scale score at 24 weeks postoperatively compared to baseline. The change value is the CGI score at 24 weeks minus the CGI score at baseline.

IPD SHARING:
Plan to Share IPD: No